CLINICAL TRIAL: NCT04176133
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Administration, Dose-Escalation Study of Entolimod on Immunosenescence in Healthy Geriatric Subjects Receiving Influenza Vaccination
Brief Title: Entolimod on Immunosenescence in Healthy Geriatric Subjects Receiving Influenza Vaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert J. Pignolo (Other)
Collaborators: Genome Protection, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Robert J. Pignolo, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-004847
Record Dates: First submitted 2019-10-30; First posted 2019-11-25 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: Vaccination; Geriatric; Immunology; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — CBLB502; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Entolimod 1 mcg (Experimental): Subjects will receive entolimod as a single dose administered intramuscularly (1mcg)
  Interventions: Drug: Entolimod; Drug: Influenza vaccine
- Entolimod 3 mcg (Experimental): Subjects will receive entolimod as a single dose administered intramuscularly (3mcg)
  Interventions: Drug: Entolimod; Drug: Influenza vaccine
- Entolimod 10 mcg (Experimental): Subjects will receive entolimod as a single dose administered intramuscularly (10mcg)
  Interventions: Drug: Entolimod; Drug: Influenza vaccine
- Placebo (Placebo Comparator): Subjects will receive a placebo as a single dose administered intramuscularly (no study drug); placebo that looks exactly like the study drug, but contains no active ingredient.
  Interventions: Drug: Placebo; Drug: Influenza vaccine

INTERVENTIONS:
Drug: Entolimod — Intramuscular (IM) single dose administration. Entolimod is provided as a sterile, clear, colorless or slightly yellow liquid for IM injection.
  Other Names: CBLB502
  Arms: Entolimod 1 mcg; Entolimod 10 mcg; Entolimod 3 mcg
Drug: Placebo — Intramuscular (IM) single dose administration, no active ingredient. A matching placebo is provided as a sterile, clear, colorless to slightly yellow liquid for IM injection in prefilled vials that are identical in appearance to the vials containing active drug.
  Arms: Placebo
Drug: Influenza vaccine — Intramuscular (IM) single dose administration. Fluzone, high-dose split virion influenza virus vaccine, Sanofi Pasteur
  Other Names: Fluzone

SUMMARY:
Researchers are evaluating the safety and effectiveness of a single administration of entolimod when administered at the same time as the influenza vaccine (flu vaccine).

ELIGIBILITY:
Inclusion:

* Men and women of age 65 years and older at the time of enrollment
* Eligible to receive Fluzone High-Dose
* Female subjects must be past menopause and not pregnant
* No history of anaphylactic reaction to gelatin, neomycin, or other vaccine component
* Must not have had the flu vaccine within the past 90 days
* Medically stable with no exacerbations or changes in medication regimen for chronic diseases in the past 3 months and no hospitalizations in the past 6 months
* Must be able to read/write English in order to provide informed consent and comply with study procedures
* Expected to be available for the duration of the study

Exclusion:

* Receipt of any other vaccines within the past 30 days prior to enrollment
* Acute illness within the last 7 days
* History of hypersensitivity to the flu vaccine or its components (including gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein).
* History of Guillain Barré syndrome (GBS)
* History of bleeding disorders
* Medical contraindication to treatment with vaccine as indicated by a history of autoimmune disease, immune deficiency, or hypersensitivity to other vaccines.
* Unstable major cardiovascular, renal, endocrine, immunological or hepatic disorder
* Systolic blood pressure (SBP) < 110 mmHg or orthostatic hypotension [>20 mmHg fall in SBP or >10 mmHg fall in diastolic blood pressure (DBP) with standing] at the time of screening.
* Evidence of an ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections) (within 14 days prior to entolimod administration). Note: Subjects with localized fungal infections of skin or nails are eligible.
* Clinical signs of febrile illness (temperature >99.5oF)
* Baseline vital signs with ≥Grade 2 abnormalities
* Significant cardiovascular disease (e.g., myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism, venous thromboembolism) within 6 months prior to study drug administration; symptomatic dysrhythmias or unstable dysrhythmias requiring medical therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; or uncontrolled Grade ≥3 hypertension (diastolic blood pressure ≥100 mmHg or systolic blood pressure ≥160 mmHg) despite antihypertensive therapy.

  o Significant screening ECG abnormalities, including unstable cardiac arrhythmia requiring medication, atrial fibrillation, 2nd-degree atrioventricular (AV) block type II, 3rd degree AV block, or Grade ≥2 bradycardia (within 14 days prior to entolimod administration).
* Inadequate hepatic function (within 14 days prior to entolimod administration):

  * Serum alanine aminotransferase (ALT) ≥3 × upper limit of normal (ULN) (Grade ≥1).
  * Serum aspartate aminotransferase (AST) ≥3 × ULN (Grade ≥1)
  * Serum alkaline phosphatase (ALP) ≥5 × ULN (Grade ≥2)
* Serum bilirubin ≥1.5 × ULN (Grade ≥1)
* Positive antiviral serology:

  * Positive hepatitis C virus (HCV) antibody or positive HCV ribonucleic acid (RNA) by quantitative PCR.
  * Positive hepatitis B surface antigen (HBsAg) and negative hepatitis B core (HBc) antibody or undetectable hepatitis B (HBV) deoxyribonucleic acid (DNA) by quantitative polymerase chain reaction (PCR) testing.
* Positive human immunodeficiency virus (HIV) antibody.
* Use of medication that might interact with the flu vaccine including (but not limited to) specifically: aminopyrine, phenytoin sodium, theophylline, and warfarin sodium.
* Any ongoing treatment with immunosuppressive or immune-stimulant therapy
* Ongoing use of systemic corticosteroids.
* Blood or blood products given within the three months prior to vaccination and two months after vaccination
* Current and/or expected receipt of chemotherapy, radiation therapy or any other cytotoxic or immunosuppressive therapy [i.e. more than 10 mg of prednisone given daily or on alternative days for 2 weeks or more in the past 3 months]
* Receipt of another investigational pharmaceutical product within 60 days of treatment
* Diagnosis of Parkinson's Disease, previous stroke, or significant cognitive impairment (defined as MMSE <20)
* Other concerns that in the opinion of the PI would preclude a subject from participating in study procedures or from completing the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pignolo, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Entolimod 1 mcg: Subjects received entolimod as a single dose administered intramuscularly (1mcg)
  Entolimod: Intramuscular (IM) single dose administration. Entolimod was provided as a sterile, clear, colorless or slightly yellow liquid for IM injection.
  Influenza vaccine: Intramuscular (IM) single dose administration. Fluzone, high-dose split virion influenza virus vaccine, Sanofi Pasteur
- Entolimod 3 mcg: Subjects received entolimod as a single dose administered intramuscularly (3mcg)
  Entolimod: Intramuscular (IM) single dose administration. Entolimod was provided as a sterile, clear, colorless or slightly yellow liquid for IM injection.
  Influenza vaccine: Intramuscular (IM) single dose administration. Fluzone, high-dose split virion influenza virus vaccine, Sanofi Pasteur
- Entolimod 10 mcg: Subjects received entolimod as a single dose administered intramuscularly (10mcg)
  Entolimod: Intramuscular (IM) single dose administration. Entolimod was provided as a sterile, clear, colorless or slightly yellow liquid for IM injection.
  Influenza vaccine: Intramuscular (IM) single dose administration. Fluzone, high-dose split virion influenza virus vaccine, Sanofi Pasteur
- Placebo: Subjects received a placebo as a single dose administered intramuscularly (no study drug); placebo that looks exactly like the study drug, but contains no active ingredient.
  Placebo: Intramuscular (IM) single dose administration, no active ingredient. A matching placebo was provided as a sterile, clear, colorless to slightly yellow liquid for IM injection in prefilled vials that are identical in appearance to the vials containing active drug.
  Influenza vaccine: Intramuscular (IM) single dose administration. Fluzone, high-dose split virion influenza virus vaccine, Sanofi Pasteur
Period: Overall Study
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Started | 20 | 19 | 6 | 16
Completed | 20 | 19 | 6 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo | Total
Number analyzed (Participants) | 20 | 19 | 6 | 16 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (6.30) | 70.7 (5.35) | 76.0 (6.78) | 73.1 (5.89) | 72.6 (6.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 3 | 6 | 29
  Male | 10 | 9 | 3 | 10 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 19 | 6 | 16 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 20 | 19 | 6 | 16 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 6 | 16 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Anti- A/H1N1 Antibody Titer
Description: Change of the anti- A/H1N1 influenza virus strains serum circulating antibodies (as assessed using hemagglutination inhibition (HAI) assay) levels from baseline to 1 month.
Time Frame: Baseline, 1 month
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
titer | 65.0 (137.23) | 73.2 (111.43) | 88.4 (123.74) | 20.3 (48.56)

2. Primary Outcome: Change in Anti-A/H3N2 Antibody Titer
Description: Change of the anti-A/H3N2 influenza virus strains serum circulating antibodies (as assessed using hemagglutination inhibition (HAI) assay) levels from baseline to 1 month.
Time Frame: Baseline, 1 month
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
titer | 58.4 (90.57) | 81.6 (138.59) | 28.0 (30.98) | 39.1 (79.84)

3. Primary Outcome: Change in Anti-B Antibody Titer
Description: Change of the anti-B influenza virus strains serum circulating antibodies (as assessed using hemagglutination inhibition (HAI) assay) levels from baseline to 1 month..
Time Frame: Baseline, 1 month
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
titer | 11.6 (18.93) | 28.3 (67.06) | 45.0 (56.48) | 10.0 (18.26)

4. Primary Outcome: Adverse Events
Description: The number of adverse events (AEs) related to dose limiting toxicities (DLTs); laboratory abnormalities; oxygen saturation and vital sign changes, and adverse electrocardiogram (ECG) findings for 1 year
Time Frame: 1 year
Measure: Number; unit: adverse event
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
adverse event | 39 | 27 | 23 | 26

5. Secondary Outcome: Time of Onset for Upper-respiratory Infections
Description: Subject self-reporting of the number of days to develop an upper-respiratory infection
Time Frame: 1 year
Population: The number of subjects to develop upper-respiratory infections were analyzed for each arm
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 10 | 9 | 2 | 3
days | 152.5 (127.4) | 302.3 (112.4) | 339.0 (0) | 157.0 (114.3)

6. Secondary Outcome: Upper Respiratory Infections
Description: The total number of subjects to self-report an upper-respiratory infection
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
Participants | 10 | 9 | 2 | 3

7. Secondary Outcome: Change in Frailty
Description: Change in self-reported 5 items frail scale. Frail scale scores range from 0-5, 1 point for each component, 0 = best 5 = worst (robust=0 points; pre-frail=0-1 points; frail 3-5 points)
Time Frame: baseline, 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
score on a scale | -0.1 (0.4) | -0.2 (0.6) | -0.2 (0.6) | 0.1 (0.5)

8. Secondary Outcome: Change in 6-minute Walk Test
Description: Distance a subject is able to walk over 6 minutes over a hard flat surface
Time Frame: baseline, 2 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
meters | 5.1 (25.64) | 11.0 (36.39) | 4.5 (9.83) | -15.8 (66.73)

9. Secondary Outcome: Change in Grip Strength
Description: Measured by a grip dynamometer as reported in units of pounds.
Time Frame: baseline, 2 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
pounds | 4.6 (17.20) | 1.1 (4.87) | 0.0 (1.79) | -0.7 (2.68)

10. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Subject's BMI calculated as weight in kilograms divided by height in meters squared. Uses measurements of height and weight obtained during study (with appropriate metric conversions)
Time Frame: baseline, 2 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
Number analyzed (Participants) | 20 | 19 | 6 | 16
kg/m^2 | 0.3 (0.58) | 0.1 (0.67) | -0.2 (0.97) | 0.1 (0.57)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for approximately 1 year for all subjects.
Arm/Group | Entolimod 1 mcg | Entolimod 3 mcg | Entolimod 10 mcg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/6 | 1/16
Other Adverse Events (participants affected / at risk) | 20/20 | 19/19 | 6/6 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entolimod 1 mcg (N=20) | Entolimod 3 mcg (N=19) | Entolimod 10 mcg (N=6) | Placebo (N=16)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entolimod 1 mcg (N=20) | Entolimod 3 mcg (N=19) | Entolimod 10 mcg (N=6) | Placebo (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 | 0 | 3 | 3
Bruising (Injury, poisoning and procedural complications) | 2 | 4 | 0 | 1
Cardiac disorders (Cardiac disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1
Dysgeusia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 1 | 0
Eye disorders (Eye disorders) | 0 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 5 | 8 | 2 | 4
Fever (General disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flu like symptoms (General disorders) | 1 | 1 | 1 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 6 | 1 | 5
Hematoma (Vascular disorders) | 2 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 3 | 1 | 0
Hemoglobinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Cardiac disorders) | 6 | 8 | 1 | 4
Hypotension (Cardiac disorders) | 1 | 3 | 3 | 1
Infections and infestations (Infections and infestations) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 13 | 9 | 3 | 5
Injury and poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Malaise (General disorders) | 1 | 2 | 0 | 2
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Nausea (General disorders) | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Respiratory and thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 1 | 0
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 2 | 4 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Wrist fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Electrocardiogram T wave abnormal (Cardiac disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04176133/Prot_SAP_000.pdf